CLINICAL TRIAL: NCT04126564
Title: Inner Engineering Online (IEO) Intervention for a Specific Company Employee Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Balachundhar Subramaniam, PI, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2019P000715
Record Dates: First submitted 2019-09-26; First posted 2019-10-15 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-08

CONDITIONS: Burnout; Stress; Depression, Anxiety
Keywords: Burnout; Stress; Anxiety; Depression; Meditation; Inner Engineering Online
MeSH Terms: conditions — Burnout, Psychological; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A cross over model ensures that both experimental and control group participants get to experience the effects of a proposed intervention. For our study, we are providing Inner Engineering Online as an intervention and both experimental and control group participants get to experience the benefits of meditation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IEO Intervention Group (Experimental): The Group 1 is the active study group which receives the online mindfulness intervention first.
  Interventions: Behavioral: Inner Engineering Online
- Control Group (Active Comparator): Group 2 will be asked to read a book or journal of their choice for first 30 days, and then recieve online mindfulness intervention (IEO).
  Interventions: Behavioral: Inner Engineering Online; Behavioral: Reading a book/ journal

INTERVENTIONS:
Behavioral: Inner Engineering Online — Inner Engineering Online (IEO) is a web based intervention administered by the Isha Foundation, a not-for-profit, global, volunteer-based organization.The Inner engineering online program is a holistic tool for promoting well-being that teaches individuals how to mindfully and effectively respond to daily stressors using yogic sciences. The program offers guided meditation and yoga practices to promote harmonizing mind-body-emotion, and energy of the individual while simultaneously promoting mindfulness, joy, and vitality. It includes seven modules of 90 minutes each, discussing meditations & yoga.
Behavioral: Reading a book/ journal — Reading a book regularly promotes knowledge enhancement, reduces stress and enhances memory among other benefits. For the purpose of this study, we advocate reading any book/ journal of participants choice routinely.
  Arms: Control Group

SUMMARY:
In this randomized controlled trial; differences in overall stress, burnout and wellbeing will be assessed for employees of a company participating in Inner Engineering Online, an online mind-body course that incorporates both meditation and yoga.

The study will be conducted in two phases, where in participants will be advised to practice meditation or read books.

DETAILED DESCRIPTION:
The benign behavioral intervention involved is Inner Engineering Online (IEO), a mind-body course that incorporates meditation and yoga, as well as reading a book or journal of their choice.The subjects will be randomized into two groups after they agree to the participate in the study. The study will be conducted in 2 phases.

Phase 1: If they are in group 1, they will participate in IEO which includes practice of meditation & yoga daily for a minimum of 30 minutes and complete a IEO activity log for 30 days.They will be asked to complete a set of questionnaires at baseline and after 30 days.If they are in group 2, they are asked to read a book or journal of their choice for 30 minutes each day for the first 30 days and complete a reading log.

Phase 2: After they complete reading for 30 days, group 2 participants will now participate in IEO which includes practice of meditation & yoga daily for a minimum of 30 minutes and complete an IEO activity log for the next 30 days. They are asked to complete a set of questionnaires at baseline, 30 days, and at 60 days.

These questionnaires aim to assess for burnout, stress, and well-being. These include:

* Maslach Burnout Inventory - Human Services Survey - 16 item questionnaire measuring burnout
* Perceived Stress Scale - 10 item questionnaire measuring stress
* Center for Epidemiology Studies depression Scale (CES-D) - 20 item questionnaire measuring depression
* Emotional Distress and Anxiety Short Form - 7 item questionnaire measuring anxiety
* Joy subscale of the Dispositional Positive Emotion Scale - 6 item questionnaire measuring happiness
* Mindful Attention Awareness Scale - 15 item questionnaire measuring mindfulness

Finally, participants of both the groups will be subjected to a 30 day follow-up surveys after a month of IEO completion. They will receive a set of previously administered questionnaire and a compliance survey at this point. Group 1 participants receive this survey at the 60 day time point while Group 2 participants receive it at 90 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age>=18 years
2. Interest in Inner Engineering Online Program

Exclusion Criteria:

1. Low English Proficiency
2. Not currently residing in United States

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2020-06-07 (Actual); Study Completion 2020-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Balachundhar Subramaniam, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Centre, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Upadhyay P, Chang TFH, Hariri S, Rallabandi S, Yathavakilla S, Novack V, Subramaniam B. The Effect of Inner Engineering Online (IEO) Program on Reducing Stress for Information Technology Professionals: A Randomized Control Study. Evid Based Complement Alternat Med. 2022 Jan 4;2022:9001828. doi: 10.1155/2022/9001828. eCollection 2022. PMID 35027938

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant were recruited from an IT firm named S2Tech. An awareness drive was conducted throughout the organization to enable participant recruitment for a period of 1 month. 82 participants were screened, 6 of whom did not meet inclusion criteria & 5 met with the exclusion criteria. All 71 participants were enrolled into the study since Aug 30 2019.
Pre-assignment Details: The 71 participants were subjected to baseline survey data collection following which they were randomized to their individual study groups.
Groups:
- Control Group Then IEO Intervention: Group 2 will be asked to read a book or journal of their choice for first 30 days, and then recieve online mindfulness intervention (IEO).
  Reading a book/ journal: Reading a book regularly promotes knowledge enhancement, reduces stress and enhances memory among other benefits. For the purpose of this study, we advocate reading any book/ journal of participants choice routinely.
  Inner Engineering Online: Inner Engineering Online (IEO) is a web based intervention administered by the Isha Foundation, a not-for-profit, global, volunteer-based organization.The Inner engineering online program is a holistic tool for promoting well-being that teaches individuals how to mindfully and effectively respond to daily stressors using yogic sciences. The program offers guided meditation and yoga practices to promote harmonizing mind-body-emotion, and energy of the individual while simultaneously promoting mindfulness, joy, and vitality. It includes seven modules of 90 minutes each, discussing meditations & yoga.
Period: Overall Study
Arm/Group | IEO Intervention Group | Control Group Then IEO Intervention
Started | 35 | 36
Study Phase I (30 Days) (1 Control participant withdrew during Study phase I) | 35 | 35
Study Phase II (30 Days) (Cross-over period where all of participants from the Control group initiated IEO intervention, 1control participant was Lost to Follow Up) | 35 | 34
Follow Up for Control Group Then IEO Intervention Group Only (30 Days) (1 participant withdrew consent from the study) | 0 | 33
Completed | 35 | 33
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- IEO Intervention Group: The Group 1 is the active study group which receives the online mindfulness intervention first.
  Phase I: Inner Engineering Online: Inner Engineering Online (IEO) is a web based intervention administered by the Isha Foundation, a not-for-profit, global, volunteer-based organization.The Inner engineering online program is a holistic tool for promoting well-being that teaches individuals how to mindfully and effectively respond to daily stressors using yogic sciences. The program offers guided meditation and yoga practices to promote harmonizing mind-body-emotion, and energy of the individual while simultaneously promoting mindfulness, joy, and vitality. It includes seven modules of 90 minutes each, discussing meditations & yoga.
- Control Group: Group 2 will be asked to read a book or journal of their choice for first 30 days, and then recieve online mindfulness intervention (IEO).
  Phase I: Reading a book/ journal: Reading a book regularly promotes knowledge enhancement, reduces stress and enhances memory among other benefits. For the purpose of this study, we advocate reading any book/ journal of participants choice routinely.
  Phase II: Inner Engineering Online: Inner Engineering Online (IEO) is a web based intervention administered by the Isha Foundation, a not-for-profit, global, volunteer-based organization.The Inner engineering online program is a holistic tool for promoting well-being that teaches individuals how to mindfully and effectively respond to daily stressors using yogic sciences. The program offers guided meditation and yoga practices to promote harmonizing mind-body-emotion, and energy of the individual while simultaneously promoting mindfulness, joy, and vitality. It includes seven modules of 90 minutes each, discussing meditations & yoga.
- Total: Total of all reporting groups
Arm/Group | IEO Intervention Group | Control Group | Total
Number analyzed (Participants) | 35 | 36 | 71
Age, Categorical [Count of Participants; unit: Participants] — Population: Of 34 participants in the Intervention arm, only 31 participants responded to the question regarding their age.
  Of 37 participants in the Control arm, only 34 participants responded to the question regarding their age.
  Participants
    number analyzed (Participants) | 31 | 34 | 65
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 31 | 34 | 65
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Of 34 participants in the Intervention arm, only 31 participants responded to the question regarding their age.
  Of 37 participants in the Control arm, only 34 participants responded to the question regarding their age.
  years
    number analyzed (Participants) | 31 | 34 | 65
    (all) | 40.5 (10.23) | 38.7 (10.19) | 39.38 (10.20)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Of 34 participants in the Intervention arm, only 31 participants responded to the question regarding their sex.
  Of 37 participants in the Control arm, only 34 participants responded to the question regarding their sex.
  Participants
    number analyzed (Participants) | 31 | 34 | 65
    Female | 17 | 16 | 33
    Male | 14 | 18 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — Population: Of 34 participants in the Intervention arm, only 31 participants responded to the question regarding their Region.
  Of 37 participants in the Control arm, only 34 participants responded to the question regarding their Region.
  Participants
    United States: number analyzed (Participants) | 31 | 34 | 65
    United States | 31 | 34 | 65

OUTCOME MEASURES:

1. Primary Outcome: Maslach Burnout Inventory Scale General Survey
Description: The study aims to evaluate changes in burnout levels affected by intervention using the Maslach Burnout Inventory scale General Survey (MBI_GS). This survey consists of 16 questions and designed for use with occupational groups other than human services and education, including those working in jobs such as customer service, maintenance, manufacturing, management, and most other professions.Sum of 16 items is reported for each study period. With possible range of total score between 0-80, a higher score indicates more burnout or worse score addressing their experience of burnout.
Time Frame: For Phase 1 analysis:Baseline to 4 weeks. For Phase 2 analysis: Baseline to 8 weeks
Population: Of 35 participants in the Intervention arm, only 34 participants responded to the question regarding their Baseline Maslach Burnout Inventory score.
  Of 36 participants in the Control arm, 1 participant withdrew from the study between 4 weeks and 8 weeks.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Control Then IEO Intervention Group: Group 2 will be asked to read a book or journal of their choice for first 30 days, and then recieve online mindfulness intervention (IEO).
  Inner Engineering Online: Inner Engineering Online (IEO) is a web based intervention administered by the Isha Foundation, a not-for-profit, global, volunteer-based organization.The Inner engineering online program is a holistic tool for promoting well-being that teaches individuals how to mindfully and effectively respond to daily stressors using yogic sciences. The program offers guided meditation and yoga practices to promote harmonizing mind-body-emotion, and energy of the individual while simultaneously promoting mindfulness, joy, and vitality. It includes seven modules of 90 minutes each, discussing meditations & yoga.
  Reading a book/ journal: Reading a book regularly promotes knowledge enhancement, reduces stress and enhances memory among other benefits. For the purpose of this study, we advocate reading any book/ journal of participants choice routinely.
Arm/Group | IEO Intervention Group | Control Then IEO Intervention Group
Number analyzed (Participants) | 35 | 36
score on a scale
  Baseline | 52 [44 to 64] | 52 [46 to 63]
  4 weeks: number analyzed (Participants) | 34 | 36
  4 weeks | 47 [37.2 to 57.2] | 47.5 [44 to 56]
  8 weeks (only for Control then IEO Intervention Group): number analyzed (Participants) | 0 | 35
  8 weeks (only for Control then IEO Intervention Group) |  | 49.5 [42 to 52.8]

2. Secondary Outcome: Perceived Stress Score Levels
Description: The study aims to evaluate changes in perceived levels of stress in survey participants and the effect Inner Engineering Online has over them. We use a validated scale for this purpose named, Perceived Stress Scale (PSS). The scale measures the degree to which situations in participant's life are appraised as stressful. This is the key secondary outcome for our study. We assess for change in perceived stress levels by analyzing the PSS score for each participant and comparing it to pre & post intervention results. PSS is a 10 question validated instrument that assesses stress. Participants are asked to rate on a scale of 0 (never) to 4 (very often) how often they agree with various statements. Items from each of the 10 questions are then summed to create a total perceived stress score, ranging of 0 to 40. The lower score indicates less stress, higher score indicates high perceived stress.
Time Frame: For Phase 1 analysis:Baseline to 4 weeks. For Phase 2 analysis: Baseline to 8 weeks
Population: Of 35 participants in the Intervention arm, 34 participants responded to the question regarding their PSS score.
  Of 36 participants in the Control arm, 1 participant withdrew from the study between 4 weeks and 8 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IEO Intervention Group | Control Group
Number analyzed (Participants) | 35 | 36
score on a scale
  Baseline | 16.9 (6.33) | 16.2 (5.65)
  4 weeks: number analyzed (Participants) | 34 | 36
  4 weeks | 13.1 (5.96) | 14.9 (5.33)
  Week 8 (only for Control Group then IEO Intervention group): number analyzed (Participants) | 0 | 35
  Week 8 (only for Control Group then IEO Intervention group) |  | 13.2 (6.81)

3. Other Pre Specified Outcome: Mindfulness Level
Description: We assess for change in Mindfulness levels by using a validated scale for this purpose namely, Mindfulness Attention Awareness Scale (MAAS). The scale measures the individuals' ability for receptive awareness and attention to present. This aids in evaluating any change on the individual's awareness levels after the Inner engineering intervention. We compute the MAAS scores for each participant which is a mean score for 15 item questionnaires and compare the pre & post intervention results to look for change. Participants are asked to rate on a scale of 1 (Almost Always) to 6 (Almost Never) to assess the frequency of occurrence of each experience. Mean is then computed using items from each of the 15 questions to create a MAAS score, ranging from 0 to 6. Higher MAAS scores indicate better mindfulness state.
Time Frame: For Phase 1 analysis:Baseline to 4 weeks. For Phase 2 analysis: Baseline to 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Group Then IEO Intervention Group: Group 2 will be asked to read a book or journal of their choice for first 30 days, and then recieve online mindfulness intervention (IEO).
  Inner Engineering Online: Inner Engineering Online (IEO) is a web based intervention administered by the Isha Foundation, a not-for-profit, global, volunteer-based organization.The Inner engineering online program is a holistic tool for promoting well-being that teaches individuals how to mindfully and effectively respond to daily stressors using yogic sciences. The program offers guided meditation and yoga practices to promote harmonizing mind-body-emotion, and energy of the individual while simultaneously promoting mindfulness, joy, and vitality. It includes seven modules of 90 minutes each, discussing meditations & yoga.
  Reading a book/ journal: Reading a book regularly promotes knowledge enhancement, reduces stress and enhances memory among other benefits. For the purpose of this study, we advocate reading any book/ journal of participants choice routinely.
Arm/Group | IEO Intervention Group | Control Group Then IEO Intervention Group
Number analyzed (Participants) | 35 | 36
score on a scale
  Baseline | 4.23 (0.92) | 4.19 (0.98)
  Week 4 | 4.64 (0.77) | 4.44 (0.81)
  Week 8 (only for Control Group then IEO Intervention group): number analyzed (Participants) | 0 | 35
  Week 8 (only for Control Group then IEO Intervention group) |  | 4.60 (0.79)

4. Other Pre Specified Outcome: Dispositional Positive Emotions Scale (DPES- Joy Subscale)
Description: We assess for change in the individuals' ability to feel joy and look for it in the mundane by using a validated scale for this purpose namely, Dispositional Positive Emotions Scale (DPES) particularly the Joy subscale. The Sub-scale measures the individuals' dispositional ability to feel joy in life. The aids in evaluating any change on the individual's joy predisposition levels after the Inner engineering intervention. We compute the DPES-JOY subscale scores for each participant which is a mean score for 6 item questionnaires and compare the pre & post intervention results to look for change. DPES-JOY scale ranges from 0 to 6 and higher DPES-JOY scale indicates higher joy in life.
Time Frame: For Phase 1 analysis:Baseline to 4 weeks. For Phase 2 analysis: Baseline to 8 weeks
Population: Of 35 participants in the Intervention arm, 34 participants responded to the question regarding their Baseline DPES- Joy subscale.
  Of 36 participants in the Control arm, 1 participant withdrew from the study between 4 weeks and 8 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IEO Intervention Group | Control Group Then IEO Intervention Group
Number analyzed (Participants) | 35 | 36
score on a scale
  Baseline | 4.22 (1.43) | 4.61 (1.19)
  Week 4 | 4.56 (1.56) | 4.64 (1.23)
  Week 8 (only for Control Group then IEO Intervention group): number analyzed (Participants) | 0 | 35
  Week 8 (only for Control Group then IEO Intervention group) |  | 4.78 (1.36)

5. Other Pre Specified Outcome: Centre for Epidemiologic Studies, Depression Scale
Description: We assess for change in the individual feeling depressed using a validated scale for this purpose namely, Centre for Epidemiologic Studies, Depression scale (CES-D). The scale comprises of 20 item questionnaires which measures the major facets of depression based on self-reported symptomatology. We compute the CES-D scale scores for each participant and compare the pre & post intervention results to look for change. Possible range of scores is 0-60 with higher scores indicating the presence of more symptomatology.
Time Frame: For Phase 1 analysis:Baseline to 4 weeks. For Phase 2 analysis: Baseline to 8 weeks
Population: Of 35 participants in the Intervention arm, only 34 participants responded to the question regarding their CES-D scores.
  Of 36 participants in the Control arm, 1 participant withdrew from the study between 4 weeks and 8 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IEO Intervention Group | Control Group
Number analyzed (Participants) | 35 | 36
score on a scale
  Baseline | 40.0 (9.07) | 40.1 (7.60)
  Week 4 | 37.2 (6.47) | 38.0 (5.97)
  Week 8 (only for Control Group then IEO Intervention group): number analyzed (Participants) | 0 | 35
  Week 8 (only for Control Group then IEO Intervention group) |  | 37.9 (5.75)

6. Other Pre Specified Outcome: Patient-Reported Outcomes Measurement Information System Emotional Distress- Anxiety Short Form Scale.
Description: We assess for change in the individual feeling anxious using a validated scale for this purpose namely, Patient-Reported Outcomes Measurement Information System (PROMIS) emotional distress- Anxiety short form scale. The scale comprises of 7 item questionnaires which measures the major facets of anxiety based on self-reported symptomatology. Sum is computed for the responses and scores range between 7-35, where higher scores indicating greater/wrose severity of anxiety. We compute the PROMIS Anxiety short form scale scores for each participant and compare the pre & post intervention results to look for change.
Time Frame: For Phase 1 analysis:Baseline to 4 weeks. For Phase 2 analysis: Baseline to 8 weeks
Population: Of 35 participants in the Intervention arm, only 34 participants responded to the question regarding their Baseline PROMIS score. Of 36 participants in the Control arm, 1 participant withdrew from the study between 4 weeks and 8 weeks.
  Of 36 participants in the Control arm, 1 participant withdrew from the study between baseline to 4 weeks, and 1 participant withdrew from the study between 4 weeks and 8 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IEO Intervention Group | Control Group Then IEO Intervention Group
Number analyzed (Participants) | 35 | 36
score on a scale
  Baseline | 16.4 (5.19) | 16.3 (4.69)
  Week 4 | 13.0 (5.62) | 14.6 (5.58)
  Week 8 (only for Control Group then IEO Intervention group): number analyzed (Participants) | 0 | 35
  Week 8 (only for Control Group then IEO Intervention group) |  | 13.0 (5.37)

ADVERSE EVENTS:
Description: Death, serious adverse events, and other (non-serious adverse events) were not assessed for this study.
Arm/Group | IEO Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Although our study has a rigorous experimental design by utilizing random assignment and active control, the study is limited by its small sample size. Future study may re-examine the effectiveness of IEO in promoting occupational health by using a larger and diverse sample.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/64/NCT04126564/Prot_SAP_000.pdf